CLINICAL TRIAL: NCT02027168
Title: Effectiveness of Manual Physical Therapy to Improve Endocrine Levels in Women
Status: Terminated | Type: Observational
Sponsor: Clear Passage Therapies, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: FSH-2012-001
Record Dates: First submitted 2014-01-02; First posted 2014-01-06 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: FSH Hypersecretion; Endocrine System Diseases; Infertility
Keywords: infertility; elevated FSH; alternative treatment; Clear Passage Approach; Clear Passage Physical Therapy
MeSH Terms: conditions — Endocrine System Diseases; Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CPA treatment: CPA treatment group receives 20 hours of patient centered manual physical therapy
  Interventions: Other: CPA

INTERVENTIONS:
Other: CPA — Site specific, patient centered manual physical therapy regimen focused on restoring function to the entire body
  Other Names: Clear Passage Approach; Wurn Technique

SUMMARY:
This study will examine the impact of manual physical therapy on endocrine function in women diagnosed as being infertile due to elevated follicle stimulating hormone (FSH) levels (10 mIU/mL or higher) on days 2-5 of their menstrual cycle. It is hypothesized that the manual physical therapy will decrease FSH levels.

DETAILED DESCRIPTION:
This study will investigate the effect of manual physical therapy on the endocrine levels of women by comparison of pre- and post- treatment hormone levels (FSH, LH and Estradiol). Secondary measures include assessment of pain and sexual function via questionnaires.

Hormones will be measured at prescribed time points:

* baseline: 30-60 days before treatment
* pre-treatment: 7-30 days before treatment
* post treatment 1: 10-30 days post treatment
* post treatment 2: 30-60 days post treatment

Pain and sexual function questionnaires will be completed:

* baseline: 30-60 days before treatment
* pre-treatment: 7-30 days before treatment
* post treatment 1: 30 days post treatment
* post treatment 2: 60 days post treatment

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as infertile
* FSH greater than 10mIU/mL on days 2-5 of menstrual cycle
* Regular menstrual cycle
* Residing in the US, accessible to a LabCorp testing facility

Exclusion Criteria:

* Active infection including HIV or inflammation
* Cancer within the past 5 years
* Currently pregnant
* Hemophilia, abnormal bleeding or clotting disorder
* Immune system disorder
* Abnormal ovarian cyst or endometrioma
* BMI of 35 or greater
* Any other condition in which deep manual physical therapy is contraindicated
* Currently taking any fertility medications or planning to take any fertility related medications during the course of the study. This includes all ovarian stimulating medications, artificial hormones and birth control medications.
* Participation in any assisted reproductive technique (such as IVF) other than intra-uterine insemination during the course of the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with elevated FSH levels that undergo the CPA treatment
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in endocrine levels post treatment | baseline, pre-treatment and 30 and 60 days post treatment
  Change in FSH, LH and estradiol levels from baseline and pre-treatment, baseline and 30 and 60 day post treatment.

SECONDARY OUTCOMES:
Pain levels and sexual function before treatment | 30 days before treatment
  Pain levels and sexual function before treatment as compared to baseline.
Pain levels and sexual function post treatment | 30 days post treatment
  Pain levels and sexual function as measured by survey 30 days post treatment compared to baseline.
Pain levels and sexual function post treatment | 60 days post treatment
  Pain levels and sexual function as measured by survey 60 days post treatment compared to baseline.
Pregnancy | study duration; 60 days post treatment
  Subjects will be monitored for natural intrauterine pregnancy for the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Wurn, LMT, Principal Investigator — Clear Passage Physical Therapy
Locations (1):
- Clear Passage Physical Therapy, Gainesville, Florida, United States

REFERENCES:
- [Background] Wurn BF, Wurn LJ, King CR, Heuer MA, Roscow AS, Hornberger K, Scharf ES. Treating fallopian tube occlusion with a manual pelvic physical therapy. Altern Ther Health Med. 2008 Jan-Feb;14(1):18-23. PMID 18251317
- [Background] Wurn LJ, Wurn BF, King CR, Roscow AS, Scharf ES, Shuster JJ. Increasing orgasm and decreasing dyspareunia by a manual physical therapy technique. MedGenMed. 2004 Dec 14;6(4):47. PMID 15775874
- [Background] Wurn BF, Wurn LJ, King CR, Heuer MA, Roscow AS, Scharf ES, Shuster JJ. Treating female infertility and improving IVF pregnancy rates with a manual physical therapy technique. MedGenMed. 2004 Jun 18;6(2):51. PMID 15266276